CLINICAL TRIAL: NCT02380963
Title: The Effect of Incorporating Soy Protein Foods in the Colorado Diet for Weight Loss and Maintenance
Brief Title: Effect of Soy Protein and Colorado Diet on Weight Loss and Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DuPont Nutrition and Health (Industry)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1152341
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Overweight; Obesity; Weight Loss
Keywords: Soy; Obesity; Weight Loss; Muscle; Cardiovascular Disease; Colorado Diet
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Cardiovascular Diseases

ARMS (2):
- Colorado Diet with soy protein (Experimental)
  Interventions: Dietary Supplement: Colorado Diet with soy protein foods.
- Colorado Diet (Active Comparator)
  Interventions: Behavioral: Colorado Diet with monetary payments

INTERVENTIONS:
Dietary Supplement: Colorado Diet with soy protein foods. — Phase 1 (week 1-2): Participants will be given soy protein powder and asked to consume 3 protein shakes per day.
  Phase 2 (week 3-8): Participants will be given both protein powder and soy patties designed to be similar to other phase 2 acceptable foods and will be asked to consume 2 soy protein shakes and 1 soy patty per day.
  Phase 3 (week 9-16): Participants will be given protein powder, soy patties, and protein bars designed to be similar to other phase 3 acceptable foods and will be asked to consume 1 soy protein shake, 1 soy patty and 1 soy protein bar per day.
  Maintenance Phase (month 5-12): Participants will continue to receive study food products (protein powder, patties and protein bars)
  Arms: Colorado Diet with soy protein
Behavioral: Colorado Diet with monetary payments — Phase 1 (week 1-2): Participants will be given monetary stipend and asked to consume 3 non-soy protein shakes per day.
  Phase 2 (week 3-8): Participants will be given monetary stipends and asked to consume 2 non-soy protein shakes per day.
  Phase 3 (week 9-16): Participants will be given monetary stipend and asked to consume 1 non-soy protein shake and 1 non-soy protein bar per day.
  Maintenance Phase (month 5-12): Participants will continue to receive monetary stipend.
  Arms: Colorado Diet

SUMMARY:
Dietary protein is a key element of most effective weight loss regimens. This study will investigate the effects of consuming soy protein on body composition and cardiometabolic health within the context of an effective weight loss and maintenance program called the Colorado Diet.

DETAILED DESCRIPTION:
This is a randomized study comparing the efficacy of inducing weight loss of two treatment arms all based on the Colorado Diet. Subjects will be randomly assigned to one of two study arms and instructed to follow the Colorado Diet by participating in weekly State of Slim group classes. Subjects will be followed in the study for one year. The Colorado Diet consists of 3 phases: phase 1 (week 1-2), phase 2 (weeks 3 - 8), and phase 3 (weeks 9 - 16). The maintenance phase lasts from months 5 - 12. Body weight will be monitored at each study visit and body composition will be determined using DXA. Blood lipid and lipoprotein concentrations, health & wellness questionnaires, and fitness measures will also be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 27-40
* Weight stable (have not lost or gained more than 10 pounds in the last 3 months)
* Generally healthy
* Able to exercise 70 minutes per day at moderate intensity
* Willing and able to participate in a State of Slim group class for the first 16 weeks of the study and willing to participate in 5 study visits over the 12 month study period.

Exclusion Criteria:

* Pregnant or trying to become pregnant.
* Diagnosis of type 1 or type 2 diabetes
* Individuals following a vegetarian only diet
* Food allergies (to soy, dairy, wheat/gluten, or peanut)
* Taking medications that could cause weight loss or weight gain or alter plasma lipids (such as steroids, tricyclic antidepressants, chemotherapy, antipsychotics, prescribed or OTC weight loss agents, statins, fibrates, niacin, etc). Oral contraceptives can be used as long as subject agrees to not change use of these during the study.
* Known renal disease
* Clinical hypothyroidism
* Current alcohol or drug abuse or dependence (Subjects who have quit smoking in the last 6 months will be excluded. Smokers whose smoking habits have been stable for the last 6 months and which remain stable during the study can be included).
* Any medical condition for which following a diet and/or 70 minutes of exercise daily would be inadvisable
* LDL cholesterol levels above 190 mg/dl or triglycerides above 400 mg/dl.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Body weight & body composition | 0, 2, 4, 8, 12 mths
  Changes in skeletal muscle mass and fat mass will be measured using dual-energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Blood lipid and lipoproteins | 0, 2, 4, 8, 12 mths
  Changes in lipids and lipoproteins will be measured using the Vertical Auto Profile (VAP) Test
C-reactive protein | 0, 2, 4, 8, 12 mths
  Changes in inflammatory status will be assessed by measuring circulating c-reactive protein
Level of Fitness | 0, 12 mths
  Changes in the level of fitness will be measured by a 3 minute step test, grip strength, and flexibility testing.
Quality of Life | 0, 4, 8, 12 mths
  Changes in the quality of life will be measured via Wellness Assessment Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: James O Hill, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Anschutz Health and Wellness Center, University of Colorado, Aurora, Colorado, United States